CLINICAL TRIAL: NCT01365039
Title: A Study to Evaluate the Safety and Efficacy of a Novel Contact Lens for Daily Disposable Use
Brief Title: Safety and Efficacy of a Contact Lens for Daily Disposable Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 690
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2013-11

CONDITIONS: Myopia
Keywords: contact lens
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test lens (Experimental): Test contact lens will be worn on a daily disposable wear basis.
  Interventions: Device: Test, daily disposable contact lens
- SofLens lens (Active Comparator): The currently marketed Bausch + Lomb SofLens daily disposable contact lens. Worn on a daily disposable wear basis.
  Interventions: Device: SofLens daily disposable contact lens

INTERVENTIONS:
Device: Test, daily disposable contact lens — Test lenses will be worn on a daily disposable wear basis. New study lenses will be dispensed at the Screening/Dispensing, 1-Month, and 2-Month Follow-up Visits in sufficient quantities to maintain a daily disposable wear modality.
  Arms: Test lens
Device: SofLens daily disposable contact lens — Control lenses will be worn on a daily disposable wear basis. New study lenses will be dispensed at the Screening/Dispensing, 1-Month, and 2-Month Follow-up Visits in sufficient quantities to maintain a daily disposable wear modality.
  Arms: SofLens lens

SUMMARY:
This study is to evaluate the safety and efficacy of a new hydrogel daily disposable contact lens compared to the Bausch + Lomb SofLens® daily disposable contact lens when worn by current soft contact lens wearers on a daily disposable wear basis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be myopic and require lens correction from -0.50 D to -6.00 D in each eye.
* Subjects must be correctable through spherocylindrical refraction to 40 logMAR letters or better (distance, high contrast) in each eye.
* Subjects must be free of any anterior segment disorders.
* Subjects must be adapted soft contact lens wearers and agree to wear their study lenses on a daily disposable wear basis for approximately 3 months.

Exclusion Criteria:

* Subjects with any systemic disease currently affecting ocular health or which in the Investigator's opinion may have an effect on ocular health during the course of the study.
* Subjects using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Subjects with any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Subjects who have had any corneal surgery (eg, refractive surgery).
* Subjects who are allergic to any component in the study care products.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Barna, CCRA, Principal Investigator — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Inc., Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 173 participants (346 eyes) were enrolled at 11 investigative sites in the United States (US), the first participant was enrolled in the study on 6/13/2011, the last participant exited the study on 10/1/2011.
Pre-assignment Details: This was a 3 month randomized, parallel, bilateral, single-masked study. One participant discontinued the study.
Groups:
- SofLens Lens: The currently marketed Bausch + Lomb SofLens daily disposable contact lens. Worn on a daily disposable wear basis.
  SofLens daily disposable contact lens : Control lenses will be worn on a daily disposable wear basis. New study lenses will be dispensed at the Screening/Dispensing, 1-Month, and 2-Month Follow-up Visits in sufficient quantities to maintain a daily disposable wear modality.
- Test Lens: Test contact lens will be worn on a daily disposable wear basis.
  Test, daily disposable contact lens : Test lenses will be worn on a daily disposable wear basis. New study lenses will be dispensed at the Screening/Dispensing, 1-Month, and 2-Month Follow-up Visits in sufficient quantities to maintain a daily disposable wear modality.
Period: Overall Study
Arm/Group | SofLens Lens | Test Lens
Started | 86 | 87
Completed | 85 | 87
Not Completed | 1 | 0
Not completed — Study related symptoms and complaints | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- SofLens: The currently marketed Bausch + Lomb SofLens daily disposable contact lens. Worn on a daily disposable wear basis.
  SofLens daily disposable contact lens : Control lenses will be worn on a daily disposable wear basis. New study lenses will be dispensed at the Screening/Dispensing, 1-Month, and 2-Month Follow-up Visits in sufficient quantities to maintain a daily disposable wear modality.
- Total: Total of all reporting groups
Arm/Group | SofLens | Test Lens | Total
Number analyzed (Participants) | 86 | 87 | 173
Age, Customized [Number; unit: participants]
  Between 18 and 40 years | 86 | 87 | 173
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 56 | 120
  Male | 22 | 31 | 53
Region of Enrollment [Number; unit: participants]
  United States | 86 | 87 | 173

OUTCOME MEASURES:

1. Primary Outcome: Slit Lamp Findings > Grade 2
Description: Statistical non-inferiority of Slit Lamp Findings > Grade 2 at any visit between the Test and Control lenses
Time Frame: 4 visits over 3 months
Population: Over All Follow-up Visits, Eyes with Findings > Grade 2 (All Dispensed Eyes)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | SofLens Lens | Test Lens
Number analyzed (Participants) | 86 | 87
Number analyzed (eyes) | 172 | 174
eyes | 0 | 1

2. Primary Outcome: High Contrast, Distance logMAR Visual Acuity (VA)
Description: Mean high contrast, distance logMAR VA for each eye between the Test and Control lenses. For each eye, logMAR VA will be averaged over all follow-up visits as the primary endpoint
Time Frame: 4 visits over 3 months
Population: All Eligible, Dispensed Eyes
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | SofLens | Test Lens
Number analyzed (Participants) | 86 | 87
Number analyzed (eyes) | 172 | 174
logMAR | -0.028 (0.040) | -0.025 (0.040)

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | SofLens Lens | Test Lens
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/87
Other Adverse Events (participants affected / at risk) | 0/86 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other